CLINICAL TRIAL: NCT02891525
Title: The Effect of Caloric and Non-caloric Sweeteners on Hunger, Gastrointestinal Hormones as Well as on Antral and Duodenal Motility
Brief Title: The Influence of Sweet Substrates on Hunger, Gastrointestinal Hormones and the Migrating Motor Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GIMotilitySweetTaste
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
MeSH Terms: interventions — Glucose; Fructose; acetosulfame

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50g glucose intragastric (Active Comparator): 50g glucose dissolved in 250mL tap water given via nasogastric tube
  Interventions: Dietary Supplement: 50g glucose
- 25g fructose intragastric (Active Comparator): 25g glucose dissolved in 250mL tap water given via nasogastric tube
  Interventions: Dietary Supplement: 25g fructose
- 220mg acesulfame-K intragastric (Active Comparator): 220mg acesulfame-K dissolved in 250mL tap water given via nasogastric tube
  Interventions: Dietary Supplement: 220mg acesulfame-K
- 250mL tap water intragastric (Placebo Comparator): 250mL tap water given via nasogastric tube
  Interventions: Dietary Supplement: 250mL tap water

INTERVENTIONS:
Dietary Supplement: 50g glucose
  Arms: 50g glucose intragastric
Dietary Supplement: 25g fructose
  Arms: 25g fructose intragastric
Dietary Supplement: 220mg acesulfame-K
  Arms: 220mg acesulfame-K intragastric
Dietary Supplement: 250mL tap water
  Arms: 250mL tap water intragastric

SUMMARY:
In this study, the investigators aimed at evaluating the role of sweet taste receptors in the gastrointestinal tract (GIT). Intragastric administration of glucose, fructose or acesulfame-K were compared with placebo administration for their effects on gastrointestinal motility, gut hormone release (motilin, ghrelin, glucagon-like peptide-1 (GLP-1) and insulin) and hunger feelings.

ELIGIBILITY:
Inclusion Criteria:

* BMI<30 kg/m² for the lean volunteers
* Female or male subjects aged 18 to 60
* Subject is capable and willing to give informed consent
* Female volunteers of child bearing potential must use oral, injected or implanted hormonal methods of contraception

Exclusion Criteria:

* Female volunteer is pregnant or breastfeeding
* GI diseases, major abdominal surgery
* Volunteers that have food allergies, especially fructose intolerance
* Major psychiatric illnesses
* Volunteers that use drugs affecting the GI tract or the central nervous system
* Volunteers suffering from an endocrine disease such as diabetes, Cushing's disease, Addison's disease, hypothalamic tumor
* Volunteers that have undergone surgical procedure for weight loss

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal motility measured by antroduodenal high-resolution manometry | 3 hours after administration, continuous measurement with high resolution manometry

SECONDARY OUTCOMES:
Change in gut hormone release measured by specific radioactive immunoassays | 3 hours after administration, blood sample every 15 min
Change in subjective hunger and satiety scores measured by visual analogue scales of 100 mm | 3 hours after administration, assessment every 5 min

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof., Principal Investigator — Universitaire Ziekenhuizen KU Leuven

REFERENCES:
- [Derived] Meyer-Gerspach AC, Biesiekierski JR, Deloose E, Clevers E, Rotondo A, Rehfeld JF, Depoortere I, Van Oudenhove L, Tack J. Effects of caloric and noncaloric sweeteners on antroduodenal motility, gastrointestinal hormone secretion and appetite-related sensations in healthy subjects. Am J Clin Nutr. 2018 May 1;107(5):707-716. doi: 10.1093/ajcn/nqy004. PMID 29722834